CLINICAL TRIAL: NCT00628797
Title: Multizenter-Studie Zur UVA-1 Therapie für Die Hautbeteiligung Bei Systemischer Sklerodermie
Brief Title: Effectiveness of UVA1-irradiation in the Treatment of Early Skin Fibrosis in Patients Suffering From Systemic Sclerosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of recruitement
Sponsor: Nicolas Hunzelmann (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor-Investigator, Nicolas Hunzelmann, Prof. Dr. N. Hunzelmann, University of Cologne
Organization: University of Cologne (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-200
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Systemic Scleroderma; Systemic Sclerosis
Keywords: systemic sclerosis; skin fibrosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Ultraviolet Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A UVA1 B no UVA1 (Other): half body irradiation with random allocation right and left; after three months of treatment treatment of both sides
  Interventions: Other: UVA1
- A UVA1 (Experimental)
  Interventions: Radiation: UVA1; Other: UVA1

INTERVENTIONS:
Radiation: UVA1 — intraindividual half body irradiation
  Other Names: ultraviolet light
  Arms: A UVA1
Other: UVA1 — 60 J/cm2 at least 36 tx
  Other Names: Ultraviolet light

SUMMARY:
Systemic scleroderma (SSc) is a rare chronic inflammatory diseae of the connective tissue involving the skin and internal organs. To date there is no proven therapy for the skin fibrosis available. A number of case reports and small uncontrolled cohort studies suggest that UVA1 therapy may improve skin fibrosis. The aim of this study is therefore to investigate whether treatment UVA1 in deed is effective in treating skin fibrosis in SSc using a randomized, intraindividual half body irradiation protocol.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis ACR criteria
* skin fibrosis at least involving the distal third of the lower arm

Exclusion Criteria:

* photosensitizing drugs
* recent UV therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
modified skin score | 3 months

SECONDARY OUTCOMES:
modified skin score | 6 months
histologic examination | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Hunzelmann, Principal Investigator — University of Cologne, Dept. of Dermatology
Locations (2):
- Germany (2):
  - University of Tuebingen, Dept. of Dermatology, Tübingen, Baden-Wurttemberg
  - University of Cologne, Dept. of Dermatology, Cologne, North Rhine-Westphalia